CLINICAL TRIAL: NCT04173299
Title: Does Early TIPS Improve Survival for Cirrhotic Patients With Acute Esophageal Variceal Bleeding Admitted in Intensive Care Unit?
Brief Title: Early TIPS in Real Life for Patient Admitted to Intensive Care Unit
Acronym: REALYTIPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Departmental Hospital Vendee (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC19_0422
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Esophageal Varicose Veins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Tips: Patients wtih early tips for Acute esophageal variceal bleeding
  Interventions: Procedure: early tips
- stantard treatment: patients with standard treatment (medical + endoscopic) for Acute esophageal variceal bleeding

INTERVENTIONS:
Procedure: early tips — patients with early tips
  Groups: Early Tips

SUMMARY:
Acute esophageal variceal bleeding (AEVB) is a serious complication of cirrhosis, with high morbidity and mortality. The latest European recommendations(1) recommend the early implementation, within 72 hours following esophageal variceal bleeding, of a transhepatic porto-systemic shunt set up by transjugular route (TIPS) called "early TIPS" in patients at high risk of recurrence, i.e. Child C<14 or Child B with active bleeding at the time of endoscopy. The implementation of early TIPS appears to improve survival without transplantation in these patients, although the benefit among Child B patients without active bleeding has yet to be demonstrated.

Renal failure is a determining factor in the prognosis of the cirrhotic patient. For patients with refractory ascites, or type 2 hepato-renal syndrome (i.e. chronic renal failure related to portal hypertension), the use of TIPS is recommended. Although a few studies with low levels of evidence have reported a benefit in the placement of TIPS in hepato-renal syndrome type 1 (i.e. acute renal failure related to portal hypertension), the European recommendations do not recommend the use of TIPS in this context due to lack of studies on the subject. Some studies have shown an improvement in renal function after performing TIPS in refractory ascites. To date, no studies have evaluated the impact of the implementation of early-TIPS on renal function in intensive care patients.

The investigators would like to evaluate the impact on survival without liver transplantation on D28 of the implementation of early-TIPS in cirrhotic patients with AEVB requiring ICU hospitalization, compared to standard treatment (medical and endoscopic).

DETAILED DESCRIPTION:
Using electronic patient data monitoring systems, the investigators reviewed all patients with a diagnosis of cirrhosis admitted to ICUs at the Nantes University Hospital, and departmental Hospital of Vendée from January 1, 2012, to december 31, 2018. For enrolled patients, general clinical characteristics were collected. Patients were categorized into two groups according to the type of treatment performed: early TIPS or standard treatment.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age >18 years) with cirrhosis Admitted in Intensive Care Unit Cirrhosis Child B or Child C With Acute esophageal variceal bleeding confirmed by endoscopy.

Exclusion Criteria:

Patients under guardianship Patients with a decision to limit care at the admission Patients with already a TIPS. Patients with a invasive multifocal hepatocellular carcinoma pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to intensive care between 2012 and 2018 for rupture of esophageal varices with cirrhosis Child C≤14 or Child B.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
survival without liver transplantation | day 28
  Comparison of survival without liver transplantation on day 28 between the two groups.

SECONDARY OUTCOMES:
day 90 mortality | Comparison of day 90 mortality between the two groups.
  Comparison of recurrence rates of Acute eosophageal variceal bleeding

IPD SHARING:
Plan to Share IPD: No